CLINICAL TRIAL: NCT02037555
Title: A Prospective, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Preoperative Antithrombin Supplementation in Patients Undergoing High-Risk Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Safety and Efficacy of Preoperative Antithrombin Supplementation in Patients Undergoing High-Risk Cardiopulmonary Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Covance (Industry); Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI1307
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
Keywords: Antithrombin; Cardiopulmonary bypass
MeSH Terms: interventions — Antithrombin III; Antithrombins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AT-III (Human) (Experimental): Single intravenous dose of AT-III (Human) sufficient to achieve an absolute increase of 20% (percentage points) above pretreatment AT levels according the following formula:
  AT-III (Human) dose (IU) required = (20) × (subject weight in kg) / 1.4
  Interventions: Biological: AT-III (Human)
- Placebo (Placebo Comparator): Single intravenous administration of placebo at a volume equivalent to the volume for the calculated AT-III (Human) dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AT-III (Human) — AT-III (Human) is an antithrombin concentrate prepared from pooled human plasma. AT-III (Human) is provided as a freeze-dried preparation for intravenous use. The AT-III (Human) preparation is reconstituted in 10 or 20 mL of sterile water for injection prior to intravenous administration.
  Other Names: Antithrombin
  Arms: AT-III (Human)
Other: Placebo — 0.9% Sodium Chloride for Injection, United States Pharmacopeia
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled study. The purpose of this study is to determine the safety and effectiveness of human-derived antithrombin III (AT-III [Human]) supplementation prior to high-risk, non-emergency, cardiac surgery with cardiopulmonary bypass (CPB). A total of 404 adult subjects undergoing CPB who meet the study eligibility criteria were planned to be randomized to receive either AT-III (Human) or placebo.

DETAILED DESCRIPTION:
The primary objective of this clinical study was to compare the percentage of subjects with any component of a 7 item major morbidity composite (postoperative mortality, stroke, acute kidney injury ([AKI]), surgical re-exploration, arterial or venous thromboembolic event, prolonged mechanical ventilation, or infection) between 2 groups of subjects randomly allocated to receive preoperative supplementation of AT-III (Human) (Antithrombin-III ([Human ]) or Placebo.

The secondary objectives of this clinical study were the following:

* To compare postoperative antithrombin III (AT) levels at the Intensive Care Unit (ICU) admission between the AT-III (Human) treatment group and Placebo control group
* To compare the following perioperative outcomes between the AT-III (Human) treatment group and Placebo control group:

  * Postoperative chest-drain blood loss in the first 12 and 24 hours after surgery
  * Transfusion requirements
  * Need for surgical re-exploration
  * Low cardiac output syndrome
  * Myocardial Infarction (MI)
  * Stroke
  * AKI
  * Arterial or venous thromboembolic events
  * Infections
  * Prolonged mechanical ventilation (>24 hours)
  * All-cause postoperative mortality
  * ICU stay duration
  * Prolonged ICU stay (>6 days)
  * Length of hospital stay

Additionally, safety objectives included the evaluation of AT III (Human) for clinical safety including adverse events (AEs), risks for bleeding, clinical laboratory testing, physical exam, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. At least 18 years of age.
3. Subject needed non-emergency cardiac surgery with CPB.
4. Types of cardiac operations permitted: complex/combined procedures (CABG+valve), double/triple valve repair/replacement, ascending aorta/aortic arch surgeries. Isolated CABG or single valve repair/replacements were allowed only if subject had received preoperative heparin >2 days.

   - Following the incorporation of Protocol Version 4.0 (Amendment 3 dated 02 Apr 2015), this criterion was revised to include complex/combined procedures (CABG+valve), double/triple valve repair/replacements, ascending aorta/aortic arch surgeries (without baseline AT level restriction or preoperative heparin requirement). OR isolated CABG or single valve repair/replacements were allowed only if either (a) AT level was less than 80% OR (b) preoperative heparin was received ([UFH for at least 12 hours; LMWH for more than 5 days).
5. Subject had a baseline AT level of less than 80%.

   * Following incorporation of Protocol Version 3.0 (Amendment 2 dated 02 Sep 2014) this was changed to Subject had a Prescreening/Screening and baseline local lab AT level of less than 80%.
   * Following the incorporation of Protocol Version 4.0 (Amendment 3 dated 02 Apr 2015) this criterion was deleted and noted as "Not applicable - intentionally left blank for data management purposes (consistency in eCRF capture of eligibility criteria historically)."
6. Subject had signed informed consent form.
7. Subject was willing to comply with all aspects of the protocol, including blood sampling, for the total duration of the study.

Exclusion Criteria:

1. Subject needed emergency surgery.
2. Subject needed heart transplantation.
3. Subject needed the use of minimally invasive surgery.
4. Subject had previous cardiac operation.
5. Subject had infective endocarditis.
6. Subject had thromboembolic events, stroke, or ST-elevated MI within 7 days of surgery.
7. Subject had cardiogenic shock at the time of surgery.
8. Subject had renal dysfunction: creatinine levels >2 mg/dL or chronic dialysis.
9. Subject had liver dysfunction: aspartate aminotransferase (AST), alanine aminotransferase (ALT) increase ≥2-fold above the upper-limit of local lab normal ranges.
10. Subject had treatment with Clopidogrel® and Ticagrelor® within 5 days before surgery, Prasugrel® within 7 days before surgery, glycoprotein IIb/IIIa receptor blockers within 24 hours of surgery.
11. Subject had treatment with new oral anticoagulants (Apixaban®, Rivaroxaban®, Dabigatran®) within 48 hours before surgery.
12. Subject had Vitamin K antagonist therapy and an international normalized ratio (INR) >1.3 on the day of surgery.
13. Subject had platelet count <120,000/μL.
14. Subject had history or suspicion of a congenital or acquired coagulation disorder.
15. Subject had history of anaphylactic reaction(s) to blood or blood components.
16. Subject had allergies to excipients in the study drug.
17. Subject had refused to receive allogenic transfusion of blood-derived products.
18. Subject had received AT treatment within the last 3 months prior to Screening Visit.
19. Subject was pregnant. Subject had participated in any another investigational study within the last 3 months prior to Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - UC Irvine, Orange, California
  - VA Medical Center - San Francisco, San Francisco, California
  - Stanford University Hospital and Clinics, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida College of Medicine, Gainesville, Florida
  - Jackson Memorial Hospital at University of Miami, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Memorial Medical Center, Springfield, Illinois
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - St. Vincent Heart Center of IN, LLC, Indianapolis, Indiana
  - Kentucky Clinic, Lexington, Kentucky
  - Tulane University Medical, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saint Luke's Hospital, Kansas City, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - CHI Health Nebraska Heart Medical Office, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - North Shore University Hospital, New Hyde Park, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Health Fargo, Fargo, North Dakota
  - Summa Health Hospital, Akron, Ohio
  - The Lindner Center for Research & Education - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital Memphis, Memphis, Tennessee
  - St. Thomas Health, Nashville, Tennessee
  - Memorial Hermann Memorial City Medical Center, Bellaire, Texas
  - Texas Heart, Houston, Texas
  - Cardiothoracic Surgical Associates, Richmond, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

REFERENCES:
- [Derived] Moront MG, Woodward MK, Essandoh MK, Avery EG, Reece TB, Brzezinski M, Spiess B, Shore-Lesserson L, Chen J, Henriquez W, Barcelo M, Despotis G, Karkouti K, Levy JH, Ranucci M, Mondou E; Clinical Thrombate Study Group. A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Preoperative Antithrombin Supplementation in Patients at Risk for Antithrombin Deficiency After Cardiac Surgery. Anesth Analg. 2022 Oct 1;135(4):757-768. doi: 10.1213/ANE.0000000000006145. Epub 2022 Jul 25. PMID 35877927

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AT-III (Human) | Placebo
Started | 213 | 212
Dosed (Reported for Safety Results) | 201 | 198
Dosed and Operated On (Reported for Efficacy Results) | 200 | 196
Completed | 190 | 191
Not Completed | 23 | 21

BASELINE CHARACTERISTICS:
Population: All Subjects Receiving Study Treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | AT-III (Human) | Placebo | Total
Number analyzed (Participants) | 201 | 198 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (10.4) | 65.5 (12.80) | 66.1 (11.66)
Age, Customized [Count of Participants; unit: Participants]
  Age Category: <65 years | 78 | 76 | 154
  Age Category: ≥65 years | 123 | 122 | 245
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 99
  Male | 150 | 150 | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 192 | 190 | 382
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 5 | 9
  White | 194 | 189 | 383
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Any Component of a Major Morbidity Composite
Description: Major morbidity composite defined as a composite of any one or more of the following:
  1. Postoperative mortality (deaths occurring within 30 days of the operation or occurring during the primary hospitalization).
  2. Stroke (clinical diagnosis of focal or global neurological deficit of abrupt onset caused by disturbance in cerebral blood supply).
  3. Acute kidney injury (increase of serum creatinine levels to >2.0 mg/dL and twice the baseline level or a new requirement for dialysis postoperatively).
  4. Surgical reexploration (return to operating room because of bleeding, tamponade, graft occlusion or other cardiac reason).
  5. Arterial or venous thromboembolic event (perioperative myocardial or mesenteric infarction, peripheral thromboembolism, acute coronary graft thrombosis, intracardiac thrombosis, deep vein thrombosis, pulmonary embolism).
  6. Prolonged mechanical ventilation (>24 hours).
  7. Infection (deep sternal-wound infection and/or bloodstream infections).
Time Frame: Up to Day 30 +/- 4 days
Population: All subjects Treated and Operated On Excluding 4 Subjects with Non-verifiable Data
Measure: Count of Participants; unit: Participants
Arm/Group | AT-III (Human) | Placebo
Number analyzed (Participants) | 198 | 194
Participants | 68 | 58

ADVERSE EVENTS:
Time Frame: Up to Day 30 +/- 4 days
Description: Four subjects included in the participant flow table are excluded from safety and efficacy reporting. These 4 subjects, 2 from each treatment group, were subtracted from the 399 "Dosed" subjects planned for safety reporting and the 396 "Dosed and Operated on" subjects planned for efficacy reporting. The final population for safety reporting was 395 (AT-III n=199 [ie, 201-2] + Placebo n=196 [ie, 198-2]), and for efficacy reporting was 392 (AT-III n=198 [ie, 200-2] + Placebo n=194 [ie, 196-2]).
Arm/Group | AT-III (Human) | Placebo
All-Cause Mortality (participants affected / at risk) | 7/199 | 4/196
Serious Adverse Events (participants affected / at risk) | 57/199 | 57/196
Other Adverse Events (participants affected / at risk) | 185/199 | 179/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT-III (Human) (N=199) | Placebo (N=196)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 4 (4) | 0 (0)
Arrhytmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 6 (7)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 4 (4)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 4 (4)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Hepatic congestion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac vein perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary arterial pressure increased (Investigations) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 5 (5)
Embolic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Decompressive craniectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Extravasation blood (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT-III (Human) (N=199) | Placebo (N=196)
Anaemia (Blood and lymphatic system disorders) | 48 (48) | 36 (36)
Coagulopathy (Blood and lymphatic system disorders) | 13 (13) | 8 (8)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 25 (25) | 32 (32)
Leukocytosis (Blood and lymphatic system disorders) | 44 (44) | 50 (50)
Thrombocytopenia (Blood and lymphatic system disorders) | 57 (57) | 64 (64)
Arrhythmia (Cardiac disorders) | 10 (10) | 8 (8)
Atrial fibrillation (Cardiac disorders) | 56 (61) | 40 (42)
Cardiogenic shock (Cardiac disorders) | 16 (16) | 18 (19)
Low cardiac output syndrome (Cardiac disorders) | 12 (12) | 10 (10)
Tachycardia (Cardiac disorders) | 10 (10) | 14 (14)
Constipation (Gastrointestinal disorders) | 33 (34) | 40 (40)
Nausea (Gastrointestinal disorders) | 33 (34) | 39 (39)
Oedema (General disorders) | 7 (7) | 11 (11)
Oedema peripheral (General disorders) | 13 (16) | 11 (11)
Urinary tract infection (Infections and infestations) | 11 (12) | 5 (5)
Anaemia postoperative (Injury, poisoning and procedural complications) | 18 (18) | 19 (19)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 7 (8) | 11 (12)
Procedural nausea (Injury, poisoning and procedural complications) | 11 (11) | 8 (8)
Procedural pain (Injury, poisoning and procedural complications) | 54 (54) | 64 (64)
Activated partial thromboplastin time prolonged (Investigations) | 11 (11) | 11 (11)
International normalised ratio increased (Investigations) | 19 (19) | 19 (19)
Myocardial necrosis marker increased (Investigations) | 6 (6) | 10 (10)
Prothrombin time prolonged (Investigations) | 16 (16) | 19 (19)
Electrolyte imbalance (Metabolism and nutrition disorders) | 11 (11) | 11 (11)
Fluid overload (Metabolism and nutrition disorders) | 12 (12) | 15 (15)
Hyperchloraemia (Metabolism and nutrition disorders) | 10 (10) | 14 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 62 (63) | 61 (61)
Hyperkalaemia (Metabolism and nutrition disorders) | 18 (18) | 11 (11)
Hypermagnesaemia (Metabolism and nutrition disorders) | 14 (14) | 14 (14)
Hypervolaemia (Metabolism and nutrition disorders) | 17 (17) | 28 (28)
Hypocalcaemia (Metabolism and nutrition disorders) | 19 (19) | 28 (28)
Hypochloraemia (Metabolism and nutrition disorders) | 9 (9) | 11 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (15) | 14 (14)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (11) | 13 (13)
Hypovolaemia (Metabolism and nutrition disorders) | 19 (19) | 14 (15)
Insomnia (Psychiatric disorders) | 6 (6) | 12 (12)
Acute kidney injury (Renal and urinary disorders) | 29 (30) | 11 (12)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 11 (11)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 43 (43) | 48 (51)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 50 (51) | 48 (50)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 11 (12)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 16 (16)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 31 (32)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (12)
Hypertension (Vascular disorders) | 15 (15) | 19 (19)
Hypotension (Vascular disorders) | 51 (52) | 58 (61)
Hypovolaemic shock (Vascular disorders) | 9 (9) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A 12-month post-study period is reserved for a joint, multi-center publication of study results. After this period, individual sites may publish results provided that the Sponsor is allowed 30 days to review any proposed publication for removal of confidential, protected, and trademarked material prior to submission with an option to delay publication up to 60 days if needed to protect its interests. The Sponsor shall retain the option to receive acknowledgment for its sponsorship of the study.

DOCUMENTS (2):
  • Study Protocol (2015-04-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT02037555/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT02037555/SAP_001.pdf